CLINICAL TRIAL: NCT02751242
Title: Identifying Diuretic Resistance in Patients With Acute Heart Failure
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Jin H. Han, Principal Investigator, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Other Study IDs: 151931
Record Dates: First submitted 2016-04-13; First posted 2016-04-26 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Heart Failure
Keywords: Diuretic Resistance; Emergency Medicine
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serial urine at 1, 2, 4, and 6 hours
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Usual Care: All patients will receive a dose of intravenous furosemide.

SUMMARY:
The study team hypothesizes patients at risk for diuretic resistance can be identified early in their Emergency Department (ED) or hospital stay by evaluating their urine sodium and potassium concentration after an initial dose of IV loop diuretic. The goal of this pilot study is to prospectively study urinary electrolyte excretion and determine patterns of diuretic responsiveness. This study would be utilized to power an interventional study which aims to study alternative methods of treating patients who are identified as having a poor response to diuretics in the ED and hospital. This would be expected to have a significant impact on a patient's hospital course, length of stay and adverse events.

DETAILED DESCRIPTION:
Most patients hospitalized with acute heart failure (AHF) respond to intravenous (IV) loop diuretic therapy, which results in symptom improvement and discharge from the hospital after a 3-5 day stay. However, up to 20% of these patients do not respond to IV loop diuretics, and are found to be "diuretic resistant". The treatment pathway for this cohort of patients is unclear. As a result, they experience significantly longer hospital lengths of stay, consume more healthcare resources, and experience an increased proportion of adverse events. Clinicians currently do not have a reliable method of predicting who will become diuretic resistant. The diagnosis is made after hospitalization, based on poor response to diuretics resulting in escalation of therapy. The standard approach to AHF therapy is to treat all patients with IV loop diuretics, not knowing who will become diuretic resistant. When diuretics are effective in promoting diuresis and natriuresis the urinary sodium rises and the urinary potassium falls. Those patients with continued low urinary sodium despite IV diuretic administration are at risk for developing diuretic resistance. Defining diuretic resistance based on urinary electrolytes before it becomes clinically apparent would facilitate an earlier change in therapy, with an aim of preventing a prolonged hospitalization.

Recently, a method to determine diuretic responsiveness based on measurements of urinary sodium in the first 6 hours after diuretic administration has been reported. This is a novel concept, and suggests the HF provider could identify poor diuretic responsiveness within 1-2 hours of diuretic administration. This study was conducted in the inpatient setting, where subjects were enrolled up to 4 days after admission. Conducting a similar ED-based study at the time of initial diuretic administration would be important to determine if early diuretic responsiveness can also be predicted using their formula for urinary sodium output. The fractional sodium excretion, (FeNa %), represents the amount of sodium excretion (mmol/time) as a percentage of filtered load [plasma sodium concentration to glomerular filtration rate]. FeNa has been used in several studies to assess diuresis in HF patients. Baseline FeNa has been shown to be reduced to less than 1% in patients with HF and a baseline FeNa of less than 0.2% is associated with diuretic resistance. Identifying effective therapies to mitigate diuretic resistance will improve symptoms, decrease hospital length of stay, conserve healthcare resources and possibly improve morbidity and mortality.

Sodium reabsorption is finely tuned in the distal portion of the nephron by the sodium-chloride cotransporter (NCC) in the distal convoluted tubule and the epithelial sodium channel (ENaC) in the collecting duct. Although only 5-10% of filtered urinary sodium typically reaches these portions of the nephron, this represents roughly 15-times the average daily dietary sodium intake. Nearly 100% of sodium is reabsorbed in the setting of sodium depletion, hypovolemia, or certain pathogenic conditions (congestive heart failure, decompensated cirrhosis). The aldosterone-sensitive collecting duct is largely responsible for this fine regulation by its ability to maximally active ENaC-dependent sodium reabsorption. Although ENaC activity and expression can be measured in vitro (patch clamp) and animal studies (micropuncture, Western blot), assessment in clinical studies is very limited due to the inability to access adequate tissue. Therefore, investigators have used the urinary sodium/potassium ratio as an index of ENaC activity. The study team has recently developed a mass spectrometric assay for urinary exosomal epithelial sodium channel (γENaC), demonstrating a 15-fold increase during low sodium diet or during aldosterone administration. This method represents a significant technical advance and provides clinical investigators a tool to measure ENaC expression in future clinical studies. The study team anticipates that a similar approach will enable clinicians to measure the expression of additional relevant transporters and channels.

ELIGIBILITY:
Inclusion Criteria:

* Adults over age 18
* Diagnosed with AHF in the ED
* Patient or surrogate provided informed consent

Exclusion Criteria:

* Systolic Blood pressure < 90 mmHg
* Intravenous diuretic administration prior to enrollment
* Allergy to furosemide and bumetanide
* Currently receiving any form of dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult ED patients diagnosed with HF
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2016-08; Primary Completion 2017-07-31 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Natriuretic responsiveness | First 6 hours of diuretic administration
  Defined by urine sodium output

SECONDARY OUTCOMES:
Formula to predict natriuretic responsiveness | 1 and 2 hours after diuretic administration
  Na output (mmol) = Estimated Glomerular Filtration Rate (eGFR) x (BSA/1.73) x (Cr serum/Cr urine) x 60 min x 2.5 hours x (Na urine/1000ml)

CONTACTS AND LOCATIONS:
Overall Officials: Jin Han, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No